CLINICAL TRIAL: NCT02429219
Title: Prospective Study of Monitoring the Alcohol Concentration in Breathing Air During Transurethral Prostate Resection of Benign Prostate Hyperplasia (BPH) Assessing the Uptake of Irrigation Fluids
Brief Title: Saline With Alcohol in TransUrethral Resection aNd Photoselective Vaporisation of the Prostate
Acronym: SATURN-P
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Magdeburg (Other)
Responsible Party: Principal Investigator, Johann J. Wendler, MD, Dr. med., University of Magdeburg
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MD-URO-00033
Record Dates: First submitted 2015-02-19; First posted 2015-04-29 (Estimated); Last update posted 2015-04-29 (Estimated); Status verified 2015-04

CONDITIONS: Benign Prostatic Hypertrophy
MeSH Terms: conditions — Prostatic Hyperplasia | interventions — Ethanol; Transurethral Resection of Prostate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Transurethral Resection (Active Comparator): Transurethral Resection of the Prostate in Saline irrigation with ethanol
  Interventions: Drug: Saline Irrigation with Ethanol; Procedure: transurethral resection of the prostate
- Photoselective vaporisation (Experimental): Photoselective vaporisation of the Prostate in Saline irrigation with ethanol
  Interventions: Drug: Saline Irrigation with Ethanol; Procedure: photoselective vaporisation of the prostate

INTERVENTIONS:
Drug: Saline Irrigation with Ethanol — Saline Irrigation with Ethanol (alcohol)
  Other Names: ethanol containinge saline irrigation fluid
Procedure: transurethral resection of the prostate — transurethral electro-resection of the prostate (TURP)
  Other Names: TURP
  Arms: Transurethral Resection
Procedure: photoselective vaporisation of the prostate — photoselective laser-vaporisation of the prostate (PVP)
  Other Names: PVP
  Arms: Photoselective vaporisation

SUMMARY:
Transurethral therapy (TURiS / PVP) of benign prostatic hyperplasia (BPH) using an ethanol-containing saline irrigating fluid, prospective detected by breath alcohol measurement.

DETAILED DESCRIPTION:
Aim was to evaluate the amount of absorbed saline irrigation fluid during transurethral therapy of benign prostatic hyperplasia (BPH). We want to differentiate two different methods of the surgical therapy: the TransUrethral Resection in Saline (TURiS) and the Photoselective Vaporisation of the Prostate (PVP). Both methods using saline irrigation. To measure the amount of absorbed saline irrigation fluid, we added pure Ethanol to the Irrigation fluid resulting in am 0,02% ethanol containing saline irrigation fluid. The conventional TransUrethral Resection of the Prostate (TUR) method is using electrolyte free irrigation. In the literature this method is well known for the occurence of the transurethral resection syndrome ("TUR syndrome"). This is caused by absorption of electrolyte-free irrigating fluid, followed by a hyponatraemic hyperhydration, and consists of symptoms from the circulatory and nervous Systems.

ELIGIBILITY:
Inclusion Criteria:

* Patients in which a TURiS or PVP to be performed

Exclusion Criteria:

* Alcoholics,
* Patients with severe hepatic impairment,
* Epilepsy,
* Existing metabolic acidosis.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2013-11; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
last breath alcohol measurement | Every 10 minutes, the breath alcohol is measured to 2 hours after the operation. Of these unnoticed, the intervention (surgery) is carried out until the end. It's all about the detection; the patient's treatment does not change.
  Measurement will be done using a breath Alcohol device (Alcomed 3011, Envitec-Wismar Inc., Germany). The unit will be mg/l.

SECONDARY OUTCOMES:
Surgical abortion with significant Absorption of irrigation fluid | Surgery will be last on average 1 hour
  If a significant amount if Irrigation fluid is absorbed (>1,5l), the procedure will be aborted

CONTACTS AND LOCATIONS:
Overall Officials: Markus Porsch, MD, Principal Investigator — Urologic Faculty University Magdeburg
Locations (1):
- Department of Urology University Hospital Otto-von-Guericke-University Magdeburg, Magdeburg, Saxony-Anhalt, Germany

REFERENCES:
- [Result] Hermanns T, Grossmann NC, Wettstein MS, Fankhauser CD, Capol JC, Poyet C, Hefermehl LJ, Zimmermann M, Sulser T, Muller A. Absorption of irrigation fluid occurs frequently during high power 532 nm laser vaporization of the prostate. J Urol. 2015 Jan;193(1):211-6. doi: 10.1016/j.juro.2014.07.117. Epub 2014 Aug 7. PMID 25108273